CLINICAL TRIAL: NCT00369876
Title: The Association Between Anorexia and the Level of Hormones, Cytokines and Neuroendocrine Peptides in Children After Burn Injury
Brief Title: Anorexia in Children With Burn Injury and the Reactions of the Immune and Endocrine Systems
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-04-3392-OB-CTIL
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Burns; Anorexia
Keywords: Burns; Anorexia; Neuropeptide; Leptin; Adiponectin; Gherlin
MeSH Terms: conditions — Burns; Anorexia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Anorexia in children with burn injury is a common phenomenon. The study is searching for the origin of the anorexia in those children. The study correlates between the level peptides of the immune and the endocrine systems and the length of the anorexia.

DETAILED DESCRIPTION:
Burn injury lead to hypermetabolic set to heal the damaged tissue.Burn healing uses high energy consumption and as consequence is highly There is a huge activation of the endocrine system and immune system resulting a proinflamtory status.

The nutrition component has an important role in the burn healing process by reducing the healing time and also in the quality of the scar tissue. It's been observed that many burn injury patients are suffering from anorexia. Since we know pro-inflammatory status modulate satiety rises the question is there a correlation between the level peptides of the immune and the endocrine systems to anorexia in children with burn injury.

Catecholamines serum concentrations rise following a burn injury. These hormones have an important role in determining the basal metabolic rate (BMR). During the healing process the levels of growth hormone (GH) and Insulin like growth factor I (IGF-1) are reduced. Previous studies show a correlation between these lower levels and Interleukins and cytokines such as Tumor Necrosis Factor (TNF) Interleukin-6 (IL-6). Additional hormones, which are relevant, are cortisol and insulin. Cortisol levels are very high after severe burn injuries for a long period. insulin sensitivity state also has an important role in the healing process.

TNFa and IL-6, which are inflammatory factors, found to have significantly elevated serum concentrations during the healing process. They are also known to be reducers to GH sensitivity and causes anorexia.

This study will show the connection between the immune and the endocrine systems to the burn healing process and anorexia by examining the level of hormones, interleukins and neuropeptide during the burn healing. our goal is to try and improve the treatment in children with burn injury by nutritional or drug intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age below 16 years
* Abilty to feed yourself during hospitalization
* Gaining consciousness during hospitalization

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10
Dates: Start 2004-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Omer bAR-yOSEF, dR., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel